CLINICAL TRIAL: NCT04030078
Title: A Central and Eastern European Survey On PEEP Titration and Alveolar Recruitment Manoeuvres During Surgery
Status: Completed | Type: Observational
Sponsor: Péterfy Sándor Hospital (Other)
Responsible Party: Principal Investigator, Dr. Zoltán Ruszkai, Head Of Department (Dept of Anaesth and Int Care), Péterfy Sándor Hospital
Other Study IDs: 30155-2/2019/EKU
Record Dates: First submitted 2019-07-13; First posted 2019-07-23 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Ventilator-Induced Lung Injury; Positive End-Expiratory Pressure; Alveolar Recruitment Manoeuvres
Keywords: PEEP; Alveolar Recruitment Manoeuvres; Survey
MeSH Terms: conditions — Ventilator-Induced Lung Injury | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Questionnaire-based survey

SUMMARY:
The aim of this questionnaire-based survey is to evaluate the routine use of individual positive end-expiratory pressure (PEEP) and regular alveolar recruitment manoeuvres (ARM) of Central and Eastern European anaesthesiologists during general anaesthesia.

DETAILED DESCRIPTION:
Lung protective mechanical ventilation (LPV) is associated with a lower incidence of postoperative pulmonary complications (PPC). The pathophysiology of ventilator-induced lung injury and the risk factors of PPCs have been widely identified, and a perioperative lung protective concept has been elaborated in the past decades. The three main basic elements of LPV are application of low tidal volumes (TV < 6mL/kg), use of optimal levels of PEEP and regular alveolar recruitment manoeuvres. Despite growing evidence recent studies indicated that the entire intraoperative LPV concept is still not widely implemented in current anaesthesia practice even in high-risk surgical patients. However the use low TV is common, either PEEP individualization, or regular ARM are usually ignored, moreover these elements were considered unnecessary or even harmful and their reason is questioned from time to time.

The aim of this questionnaire-based survey (using Google Forms) is to evaluate the routine use of individual PEEP and regular ARM of Central and Eastern European anaesthesiologists during general anaesthesia, and will take approximately 10 minutes to complete.

The questionnaire consists of 29 mandatory-to-answer multiple and single choice questions. The first part of the form includes questions about demographics and hospital characteristics. The second part contains questions on the use of individual PEEP titration procedures and the third part includes questions about the use of alveolar recruitment manoeuvres during general anaesthesia.

An invitation letter will be sent to the national associations of anaesthesia of Croatia, Czech Republic, Hungary, Poland, Romania, Serbia and Slovakia. Answers will be collected in Google Forms spreadsheets and will be analyzed using MedCalc Statistical Software (MedCalc Software bvba, Ostend, Belgium).

Participation in this study is entirely voluntary and anonymous. Neither sensitive personal data nor contact information will be collected during the research. There are no known risks associated with this research study; however, as with any online related activity the risk of a breach is always possible.

This research does not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors, and the investigators declare that they do not have any conflict of interest with the work.

This international survey study and questionnaire was approved by Hungarian Medical Research Council (approval nr. 30155-2/2019/EKU, date 01/07/2019).

ELIGIBILITY:
Inclusion Criteria:

- All anaesthesiologists accepting to participate the survey

Exclusion Criteria:

- None

Min Age: 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Resident doctors, specialist candidates and specialist working in the field of anaesthesia, employed in Croatia, Czech Republic, Hungary, Poland, Romania, Serbia and Slovakia
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Individual PEEP | Up to 2 months, from August to September in the year 2019
  Answers of anaesthesiologists regarding the use of individual PEEP in routine anaesthetic care during general anaesthesia by completing the survey questionnaire. Multiple and single choice answers.
  Data will be expressed as percentage of respondents. Territorial and institutional differences and differences between the practice of resident doctors and specialists - if there is any - will be evaluated.
Alveolar recruitment manoeuvres | Up to 2 months, from August to September in the year 2019
  Answers of anaesthesiologists regarding the use of alveolar recruitment manoeuvres in routine anaesthetic care during general anaesthesia by completing the survey questionnaire. Multiple and single choice answers.
  Data will be expressed as percentage of respondents. Territorial and institutional differences and differences between the practice of resident doctors and specialists - if there is any - will be evaluated.

SECONDARY OUTCOMES:
Practices and preferences of PEEP titration procedures | Up to 2 months, from August to September in the year 2019
  Commonly used PEEP titration procedures during routine anaesthetic care will be evaluated by collection of answers to the survey. Data will be expressed as percentage of respondents.
Practices and preferences of alveolar recruitment manoeuvres | Up to 2 months, from August to September in the year 2019
  Commonly used methods of alveolar recruitment manoeuvres during routine anaesthetic care will be evaluated by collection of answers to the survey. Data will be expressed as percentage of respondents.
Adverse effects of alveolar recruitment manoeuvres | Up to 2 months, from August to September in the year 2019
  The most commonly observed side effects of alveolar recruitment manoeuvres will be evaluated by collection of answers to the survey. Data will be expressed as percentage of respondents.
Contraindications of alveolar recruitment manoeuvres | Up to 2 months, from August to September in the year 2019
  Opinion responses of survey participants about the contraindications of the use of any type of alveolar recruitment manoeuvres in their daily practice. Data will be expressed as percentage of respondents.

OTHER OUTCOMES:
Protocols on perioperative lung protective ventilatory management | Up to 2 months, from August to September in the year 2019
  Answers of respondents regarding the availability of written institutional protocols on perioperative lung protective ventilatory management by completing the survey questionnaire. Data will be expressed as percentage of respondents.

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Ruszkai, MD, Principal Investigator — Péterfy Hospital
Locations (1):
- Péterfy Sándor Hospital, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- See also: Survey Questionaire — https://forms.gle/Si1hFaDPh6dCPuDM8